CLINICAL TRIAL: NCT01958320
Title: Early Treatment Versus Delayed Conservative Treatment of the Patent Ductus Arteriosus in Preterm infants-a Multicenter Trial
Brief Title: Early Treatment Versus Delayed Conservative Treatment of the Patent Ductus Arteriosus
Acronym: PDA:TOLERATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC4
Record Dates: First submitted 2013-10-04; First posted 2013-10-09 (Estimated); Results first posted 2018-11-30 (Actual); Last update posted 2018-11-30 (Actual); Status verified 2018-11

CONDITIONS: Patent Ductus Arteriosus; Surgery; Necrotizing Enterocolitis; Intestinal Perforation
Keywords: patent ductus arteriosus; patent ductus arteriosus ligation; necrotizing enterocolitis; spontaneous intestinal perforation
MeSH Terms: conditions — Ductus Arteriosus, Patent; Enterocolitis, Necrotizing; Intestinal Perforation | interventions — Anti-Inflammatory Agents, Non-Steroidal

STUDY DESIGN:
Intervention Model Description: Early routine, mandated PDA treatment versus Conservative treatment only if Rescue criteria are met
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Early treatment (Experimental): Infants randomized to the early treatment group will receive "pharmacologic treatment of the PDA" to produce PDA closure. Within 24-36 hr following the last treatment dose an echocardiogram will be obtained to document the degree of ductus closure or patency.
  Echocardiograms will be obtained at 1) 10-14 days after study entry (if the PDA was open and of moderate size on the last echocardiogram), and 2) at the time of hospital discharge (if the PDA was open (any size) on the last echocardiogram). The echocardiogram obtained at discharge will be used to determine the need for outpatient follow-up.
  Interventions: Other: pharmacologic treatment of the PDA; Drug: NSAID
- Conservative Treatment (Active Comparator): Infants randomized to the Conservative Treatment approach will receive "no pharmacologic treatment of the PDA" but will be followed to determine if they meet criteria for later PDA "rescue treatment" (Infants will be eligible for rescue treatment of their persistent PDA if they meet the rescue treatment criteria.)
  Echocardiograms will be obtained at 1) 10-14 days after study entry (if the PDA was open and of moderate size on the last echocardiogram), and 2) at the time of hospital discharge (if the PDA was open (any size) on the last echocardiogram). The echocardiogram obtained at discharge will be used to determine the need for outpatient follow-up.
  Interventions: Other: no pharmacologic treatment of the PDA; Drug: NSAID

INTERVENTIONS:
Other: pharmacologic treatment of the PDA — Following randomization, infants will be treated with medications used to produce PDA closure.
  Arms: Early treatment
Other: no pharmacologic treatment of the PDA — Following randomization, infants will NOT be treated with medications used to produce PDA closure (unless they develop rescue criteria at a later point in time).
  Arms: Conservative Treatment
Drug: NSAID — Indomethacin, ibuprofen or acetaminophen will be used as standard of care treatment

SUMMARY:
The primary goal of the trial is to compare two different Patent Ductus Arteriosus (PDA) treatment approaches: 1) an "early treatment" approach or 2) a "conservative" approach. For the purposes of the study infants will be enrolled if they are delivered before 28 weeks gestation and have a moderate/large PDA present at 5-7 days after birth.

The hypothesis is: treatment of a moderate size patent ductus arteriosus (PDA) will decrease the time needed for assisted respiratory support, diuretic therapy, and gavage feeding assistance, in addition to decreasing the incidence of ductus ligations or need for future outpatient cardiology follow-up appointments. The investigators hypothesize that one or more of these benefits will occur without an increase in the time taken to achieve full enteral feedings or in the incidence of necrotizing enterocolitis (NEC) or spontaneous intestinal perforations (SIP).The investigators will be comparing the effectiveness of early pharmacologic treatment with a control group of conservatively managed infants who will only receive treatment if they meet specific criteria for "rescue treatment".

DETAILED DESCRIPTION:
Prior studies showed that, if a moderate/large Patent Ductus Arteriosus (PDA) is still present at 5 days after birth (among infants delivered at 23 and 0/7 to 25 and 6/7 weeks gestation) or at 7 days after birth (among infants delivered at 26 and 0/7 to 27 and 6/7 weeks gestation), it will persist for at least another 4-12 weeks if it is left untreated.

ELIGIBILITY:
Inclusion Criteria:

This will be a prospective randomized, multi-center, controlled trial that will enroll infants delivered between 23 & 0/7 - 27 & 6/7 weeks gestation:

1. infants must be between 5-14 days old (if delivered between 23 and 0/7 - 25 and 6/7 weeks) or 7-14 days old (if delivered between 26 & 0/7 - 27 & 6/7 weeks) and
2. have a "moderate size PDA" (defined as a PDA on echocardiogram that has at least one of the following criteria: internal ductus diameter ≥1.5 mm/kg (or PDA:LPA ratio ≥0.5), ductus flow velocity ≤2.5 m/s or mean pressure gradient across the ductus <8 mm, LA/Ao ratio ≥1.5, left pulmonary artery diastolic (or mean) flow velocity >0.2 (or >0.42) m/sec, respectively, and/or reversed diastolic flow in the descending aorta)(13, 68, 69) and
3. are receiving respiratory support consisting of either mechanical ventilation, nasal CPAP, SiPAP, or nasal cannula flow ≥2 L/min.

   -

   Exclusion Criteria:

   prior treatment with indomethacin, ibuprofen, or acetaminophen, contraindications for the use of indomethacin, ibuprofen, or acetaminophen (these include: hydrocortisone administration within 24 hrs, urine output < 1 ml/kg/h during the preceding 8 h, serum creatinine level >1.6 mg/dl, platelet count <50, 000/mm3, abnormal coagulation studies, or total bilirubin concentration (in mg/dL) > 8 x weight (in kg)), chromosomal anomalies, congenital or acquired gastrointestinal anomalies, prior episode of necrotizing enterocolitis or intestinal perforation.

   -

Ages: 5 Days to 14 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 202 (Actual)
Dates: Start 2013-12; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Clyman, MD, Principal Investigator — University of California, San Francisco
Locations (18):
- United States (13):
  - University of California San Diego, San Diego, California
  - Sharp Mary Birch Hospital for Women and Newborns, San Diego, California
  - University of California San Francisco, San Francisco, California
  - Mednax Neonatology of San Jose/Pediatrix Medical Group, San Jose, California
  - Kaiser Permanente Santa Clara, Santa Clara, California
  - South Miami Hospital, Miami, Florida
  - University of Chicago Medicine, Chicago, Illinois
  - Northshore University Health System, Evanston, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Mayo Clinic, Rochester, Minnesota
  - Morristown Medical Center, Morristown, New Jersey
  - Columbia University, New York, New York
  - Providence St Vincent Medical Center, Portland, Oregon
- University Hospital, Umea, Sweden, Umeå, Sweden
- Turkey (Türkiye) (3):
  - Ankara University School of Medicine Children's Hospital, Ankara
  - Sisli Hamidiye Etfal Training and Research Hospital, Istanbul
  - Inonu University School of Medicine Turgut Ozal Medical Center, Malatya
- University of Glasgow, Royal Hospital for Sick Children, Glasgow, Scotland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
What data in particular will be shared? Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
  What other documents will be available? Study Protocol
  When will data be available (start and end dates)? Beginning 9 months and ending 36 months following article publication.
  With whom? Researchers who provide a methodologically sound proposal.
  For what types of analyses? To achieve aims in the approved proposal.
  Proposals should be directed to clymanr@ucsf.edu. To gain access, data requestors will need to sign a data access agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Researchers who provide a methodologically sound proposal. o achieve aims in the approved proposal. Proposals should be directed to clymanr@ucsf.edu. To gain access, data requestors will need to sign a data access agreement.

REFERENCES:
- [Result] Clyman RI, Liebowitz M, Kaempf J, Erdeve O, Bulbul A, Hakansson S, Lindqvist J, Farooqi A, Katheria A, Sauberan J, Singh J, Nelson K, Wickremasinghe A, Dong L, Hassinger DC, Aucott SW, Hayashi M, Heuchan AM, Carey WA, Derrick M, Fernandez E, Sankar M, Leone T, Perez J, Serize A; PDA-TOLERATE (PDA: TO LEave it alone or Respond And Treat Early) Trial Investigators. PDA-TOLERATE Trial: An Exploratory Randomized Controlled Trial of Treatment of Moderate-to-Large Patent Ductus Arteriosus at 1 Week of Age. J Pediatr. 2019 Feb;205:41-48.e6. doi: 10.1016/j.jpeds.2018.09.012. Epub 2018 Oct 16. PMID 30340932
- [Derived] Liebowitz M, Katheria A, Sauberan J, Singh J, Nelson K, Hassinger DC, Aucott SW, Kaempf J, Kimball A, Fernandez E, Carey WA, Perez J, Serize A, Wickremasinghe A, Dong L, Derrick M, Wolf IS, Heuchan AM, Sankar M, Bulbul A, Clyman RI; PDA-TOLERATE (PDA: TOLEave it alone or Respond And Treat Early) Trial Investigators. Lack of Equipoise in the PDA-TOLERATE Trial: A Comparison of Eligible Infants Enrolled in the Trial and Those Treated Outside the Trial. J Pediatr. 2019 Oct;213:222-226.e2. doi: 10.1016/j.jpeds.2019.05.049. Epub 2019 Jun 27. PMID 31255386
- [Derived] Liebowitz M, Kaempf J, Erdeve O, Bulbul A, Hakansson S, Lindqvist J, Farooqi A, Katheria A, Sauberan J, Singh J, Nelson K, Wickremasinghe A, Dong L, Hassinger DC, Aucott SW, Hayashi M, Heuchan AM, Carey WA, Derrick M, Wolf IS, Kimball A, Sankar M, Leone T, Perez J, Serize A, Clyman RI. Comparative effectiveness of drugs used to constrict the patent ductus arteriosus: a secondary analysis of the PDA-TOLERATE trial (NCT01958320). J Perinatol. 2019 May;39(5):599-607. doi: 10.1038/s41372-019-0347-4. Epub 2019 Mar 8. PMID 30850756

RESULTS

PARTICIPANT FLOW:
Groups:
- Early Treatment: Infants randomized to the early treatment group will receive "pharmacologic treatment of the PDA" to produce PDA closure. Within 24-36 hr following the last treatment dose an echocardiogram will be obtained to document the degree of ductus closure or patency.
  Echocardiograms will be obtained at 1) 10-14 days after study entry (if the PDA was open and of moderate size on the last echocardiogram), and 2) at the time of hospital discharge (if the PDA was open (any size) on the last echocardiogram). The echocardiogram obtained at discharge will be used to determine the need for outpatient follow-up.
  pharmacologic treatment of the PDA: Following randomization, infants will be treated with medications used to produce PDA closure.
- Conservative Treatment: Infants randomized to the Conservative Treatment approach will receive "no pharmacologic treatment of the PDA" but will be followed to determine if they meet criteria for later PDA "rescue treatment" (Infants will be eligible for rescue treatment of their persistent PDA if they meet the rescue treatment criteria.)
  Echocardiograms will be obtained at 1) 10-14 days after study entry (if the PDA was open and of moderate size on the last echocardiogram), and 2) at the time of hospital discharge (if the PDA was open (any size) on the last echocardiogram). The echocardiogram obtained at discharge will be used to determine the need for outpatient follow-up.
  no pharmacologic treatment of the PDA: Following randomization, infants will NOT be treated with medications used to produce PDA closure (unless they develop rescue criteria at a later point in time).
Period: Overall Study
Arm/Group | Early Treatment | Conservative Treatment
Started | 104 | 98
Completed | 104 | 98
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Early Treatment | Conservative Treatment | Total
Number analyzed (Participants) | 104 | 98 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 104 | 98 | 202
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days after birth] — days after birth
  days after birth | 8.1 (2.1) | 8.3 (2.3) | 8.2 (2.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 55 | 111
  Male | 48 | 43 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 25 | 19 | 44
  Not Hispanic or Latino | 79 | 79 | 158
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 12 | 14 | 26
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 14 | 11 | 25
  White | 76 | 73 | 149
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 7 | 7 | 14
  Turkey | 14 | 15 | 29
  United States | 80 | 72 | 152
  United Kingdom | 3 | 4 | 7
Gestation [Mean (Standard Deviation); unit: weeks of gestation] — weeks of gestation
  weeks of gestation | 25.7 (1.2) | 25.9 (1.1) | 25.8 (1.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Infants Who Undergo in Hospital PDA Ligations or Who Have an Open Ductus at the Time of Discharge (That Need Future Outpatient Cardiology Follow-up Visits)
Description: Number of infants who undergo in hospital PDA ligations or who have an open ductus at the time of discharge (that need future outpatient cardiology follow-up visits)
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Groups:
- Early Treatment: Infants randomized to the early treatment group will receive "pharmacologic treatment of the PDA" to produce PDA closure.
  pharmacologic treatment of the PDA: Following randomization, infants will be treated with medications used to produce PDA closure.
- Conservative Treatment: Infants randomized to the Conservative Treatment approach will receive "no pharmacologic treatment of the PDA" but will be followed to determine if they meet criteria for later PDA "rescue treatment" (Infants will be eligible for rescue treatment of their persistent PDA if they meet the rescue treatment criteria.)
  no pharmacologic treatment of the PDA: Following randomization, infants will NOT be treated with medications used to produce PDA closure (unless they develop rescue criteria at a later point in time).
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 33 | 38

2. Secondary Outcome: Duration of Gavage Feeding Assistance
Description: duration of gavage feeding assistance
Time Frame: up to 20 weeks of age
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
days | 76 [66 to 104] | 80 [61 to 97]

3. Secondary Outcome: Incidence of Necrotizing Enterocolitis or Spontaneous Perforation
Description: incidence of necrotizing enterocolitis or spontaneous perforation
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 17 | 19

4. Secondary Outcome: the Average Daily Weight Gain
Description: the average daily weight gain
Time Frame: up to 20 weeks of age
Measure: Mean (Standard Deviation); unit: gm/kg/day
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
gm/kg/day | 22.5 (4.8) | 22.8 (4.6)

5. Secondary Outcome: Incidence of Bronchopulmonary Dysplasia or Death
Description: incidence of bronchopulmonary dysplasia or death
Time Frame: determined between 36-37 weeks corrected age
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 60 | 56

6. Secondary Outcome: Incidence of Death
Description: incidence of death
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 20 | 10

7. Secondary Outcome: the Incidence of Persistent Moderate-to-large PDA Shunt 10 Days After Enrollment
Description: the incidence of persistent moderate-to-large PDA shunt 10 days after enrollment The echocardiographic studies included two dimensional imaging, M-mode, color flow mapping and Doppler interrogation as previously described. A moderate-to-large PDA was defined by a ductus internal diameter ≥ 1.5mm (or PDA:left pulmonary artery diameter ratio ≥0.5) and one or more of the following echocardiographic criteria: a) left atrium-to-aortic root (LA/Ao) ratio ≥1.6, b) ductus flow velocity ≤2.5m/sec or mean pressure gradient across the ductus ≤8mm, c) left pulmonary artery diastolic flow velocity > 0.2 m/sec, and/or d) reversed diastolic flow in the descending aorta. Ductus that failed to meet these criteria were considered to be "constricted" (small or closed) and not eligible for enrollment or treatment.
Time Frame: 10 days after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 43 | 78

8. Secondary Outcome: the Incidence of Rescue Treatment Eligibility Criteria Met
Description: Infants were eligible for rescue PDA drug treatment if they met one or more of the following prespecified "Rescue" criteria: 1) Inotrope-dependent hypotension for at least 3 days. 2) Oliguria that persisted for at least 2 days with no obvious cause, other than the moderate PDA, to explain the condition. 3) Requirement for gavage feedings beyond 35 weeks corrected age due to increased work of breathing. 4) Respiratory support needed after the following postnatal ages that surpassed specific minimal ventilation and FiO2 requirements: >15 days (if still required intubation and FiO2 >0.30), >20 days (if still required intubation and FiO2 ≤0.30; or still required Nasal CPAP or Nasal ventilation and FiO2 >0.30), >30 days (if still required Nasal CPAP or Nasal ventilation and FiO2 0.25-0.30), and >45 days (if still required Nasal CPAP or Nasal ventilation and FiO2 <0.25).
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 32 | 61

9. Secondary Outcome: Number of Infants Receiving ≥ 14 Days of Diuretic Treatment
Description: number of infants receiving ≥ 14 days of diuretic treatment
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 36 | 45

10. Other Pre Specified Outcome: Number of Infants Who Received Dopamine for ≥3 Days
Description: number of infants who received dopamine for ≥3 days
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 14 | 25

11. Other Pre Specified Outcome: Incidence of Bacteremia
Description: incidence of bacteremia
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 31 | 21

12. Other Pre Specified Outcome: Incidence of Pulmonary Hemorrhage
Description: incidence of pulmonary hemorrhage
Time Frame: through hospital discharge (approximately 6 months unless death occurs first)
Measure: Count of Participants; unit: Participants
Arm/Group | Early Treatment | Conservative Treatment
Number analyzed (Participants) | 104 | 98
Participants | 2 | 2

ADVERSE EVENTS:
Time Frame: until hospital discharge (approximately 6 months unless death occurs first)
Description: The definition of serious adverse event in this trial only included the following: Necrotizing enterocolitis and death.
Arm/Group | Early Treatment | Conservative Treatment
All-Cause Mortality (participants affected / at risk) | 20/104 | 10/98
Serious Adverse Events (participants affected / at risk) | 17/104 | 19/98
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Early Treatment (N=104) | Conservative Treatment (N=98)
necrotizing enterocolitis (Gastrointestinal disorders) | 17 | 19 — NEC

LIMITATIONS AND CAVEATS:
See detailed limitations in published manuscript

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-06-19): https://cdn.clinicaltrials.gov/large-docs/20/NCT01958320/Prot_SAP_000.pdf